CLINICAL TRIAL: NCT05163808
Title: A Randomized, Double-blind, Placebo-controlled, Two-Part Study of BPN14770 in Male Adolescents (Aged 9 to < 18 Years) With Fragile X Syndrome
Brief Title: A Randomized Study of BPN14770 in Male Adolescents (Aged 9 to < 18 Years) With Fragile X Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tetra Discovery Partners (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BPN14770-CNS-204
Record Dates: First submitted 2021-12-15; First posted 2021-12-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome | interventions — BPN14770

STUDY DESIGN:
Intervention Model Description: 2 treatment Groups (Study Drug and Placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Drug (Active Comparator): Subjects will receive 15 mg BID or 25mg BID dose of BPN14770
  Interventions: Drug: zatolmilast
- Placebo Arm (Placebo Comparator): Subjects will receive matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: zatolmilast — Subjects will receive a 15 mg or 25 mg dose of zatolmilast (BPN14770) or placebo
  Other Names: BPN14770
  Arms: Study Drug
Drug: Placebo — Placebo
  Arms: Placebo Arm

SUMMARY:
This is a 2-part study, with each part having a unique set of objectives for male adolescents aged 9 to < 18 years with fragile X syndrome (FXS). Part 1 is an open-label, single-dose, pharmacokinetics (PK) assessment of BPN14770 25 mg and 50 mg, while Part 2 is double-blind (DB) and randomized between two treatment groups (Study Drug and Placebo).

DETAILED DESCRIPTION:
In amendment 4 the enrollment age range what changed to allow enrollment in participants as young as 9 years of age. This only affects Part 2 as Part 1 was completed prior to this amendment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient is male adolescent aged 9 to < 18 years. 2. Patient has FXS with a molecular genetic confirmation of the full fragile X mental retardation-1 (FMR1) mutation (≥ 200 CGG repetitions).

  3. Current treatment with ≤ 3 prescribed psychotropic medications. Anti-epileptic medications are permitted and are not counted as psychotropic medications if they are used for treatment of seizures. Anti-epileptics for other indications, such as the treatment of mood disorders, count towards the limit of permitted medications. If the subject is on 3 prescribed psychoactive medications and, in addition, is taking either a psychoactive over-the-counter medication (eg, melatonin, Benadryl, etc.) or CBD products, the investigator is encouraged to discuss eligibility with the medical monitor.

  4. Permitted concomitant psychotropic medications must be at a stable dose and dosing regimen for at least 4 weeks before screening and must remain stable during the period between screening and the commencement of study drug. Every effort should be made to keep dosing stable throughout the study.

  5. Anti-epileptic medications must be at a stable dose and dosing regimen for 12 weeks before screening and must remain stable during the period between screening and the commencement of study drug. Every effort should be made to keep dosing stable throughout the study.

  6. Patients with a history of seizure disorder who are currently receiving treatment with anti-epileptics must have been seizure-free for 3 months before screening or must be seizure-free for 2 years if not currently receiving anti-epileptics.

  7. Behavioral and other non-pharmacological treatments/interventions must be stable for 4 weeks before screening and must remain stable during the period between screening and the commencement of study drug, and throughout the study. Minor changes in hours or times of therapy that are not considered clinically significant will not be exclusionary. Changes in therapies provided through a school program, due to school vacations, are allowed.

  8. Patient must be willing to practice barrier methods of contraception while on study, if sexually active. Abstinence is also considered a reasonable form of birth control in this study population.

  9. Patient has a parent(s), legal authorized guardian(s), or consistent caregiver(s).

  10. Patient and caregiver are able to attend the clinic regularly and reliably. 11. Patient's parent(s), legal authorized guardian(s), or consistent caregiver(s) is able to understand and sign an informed consent form to participate in the study.

  12. Patient must provide assent for participation in the study if the patient has the cognitive ability to provide assent.

  13. To participate in the Part 1 PK only: subjects must be able to swallow capsules.

Exclusion Criteria:

Diagnosis and main criteria for inclusion:

The eligibility criteria are the same for all parts of the study except for Part 1 (PK), where patients must be able to swallow capsules and must weigh at least 75 lbs (34 kg) to receive the 50 mg dose.

Patient Inclusion Criteria

1. Patient is male adolescent aged 12 to < 18 years.
2. Patient has FXS with a molecular genetic confirmation of the full fragile X mental retardation-1 (FMR1) mutation (≥ 200 CGG repetitions).
3. Current treatment with ≤ 3 prescribed psychotropic medications. Anti-epileptic medications are permitted and are not counted as psychotropic medications if they are used for treatment of seizures. Anti-epileptics for other indications, such as the treatment of mood disorders, count towards the limit of permitted medications.
4. Permitted concomitant psychotropic medications must be at a stable dose and dosing regimen for at least 4 weeks before screening and must remain stable during the period between screening and the commencement of study drug.
5. Anti-epileptic medications must be at a stable dose and dosing regimen for 12 weeks before screening and must remain stable during the period between screening and the commencement of study drug.
6. Patients with a history of seizure disorder who are currently receiving treatment with anti-epileptics must have been seizure-free for 3 months before screening or must be seizure-free for 2 years if not currently receiving anti-epileptics.
7. Behavioral and other non-pharmacological treatments/interventions must be stable for 4 weeks before screening and must remain stable during the period between screening and the commencement of study drug, and throughout the study. Minor changes in hours or times of therapy that are not considered clinically significant will not be exclusionary. Changes in therapies provided through a school program, due to school vacations, are allowed.
8. Patient must be willing to practice barrier methods of contraception while on study, if sexually active. Abstinence is also considered a reasonable form of birth control in this study population.
9. Patient has a parent(s), legal authorized guardian(s), or consistent caregiver(s).
10. Patient and caregiver are able to attend the clinic regularly and reliably.
11. Patient's parent(s), legal authorized guardian(s), or consistent caregiver(s) is able to understand and sign an informed consent form to participate in the study.
12. Patient must provide assent for participation in the study if the patient has the cognitive ability to provide assent.
13. To participate in the Part 1 PK only: patients must be able to swallow capsules.

Patient Exclusion Criteria

1. Inability to successfully complete the NIH-TCB picture vocabulary and oral reading assessments at screening and baseline for Part 2 (DB). Patient must be able to complete these assessments at baseline to be randomized into Part 2; care should be taken that a patient enrolled into Part 1 (PK) possesses this ability if their desire is to continue to Part 2. The ability to complete the NIH-TBC oral reading and picture vocabulary subtest at baseline is defined as the ability to complete both subtests, with (1) confirmation from the clinician administering that the test administrations are valid (noted on the administration form), and (2) generation of valid test scores for each test.
2. History of, or current cardiovascular, renal, hepatic, respiratory, gastrointestinal, psychiatric, neurologic, cerebrovascular, or other systemic disease that would place the patient at risk or potentially interfere with the interpretation of the safety, tolerability, or efficacy of the study drug.

   • Common conditions such as mild hypertension, etc. are allowed per the PI's judgment as long as they are stable and controlled by medical therapy that is constant for at least 4 weeks before randomization.
3. Renal impairment, defined as serum creatinine > 1.25 × ULN at screening.
4. Cirrhosis, unstable chronic liver disease or acute liver disease. Hepatic impairment, defined as alanine aminotransferase or aspartate aminotransferase elevation > 2 × ULN at screening. Note: liver function tests may be repeated after 1 week to evaluate return to acceptable limits; if liver function tests remain elevated, patient is ineligible to participate. Subjects with stable chronic hepatitis B on oral anti-viral therapy and subjects cured of chronic hepatitis C may be allowed. Subjects with Gilbert syndrome are allowed.
5. Clinically significant abnormalities, in the PI's judgment, in safety laboratory tests, vital signs, or 12-lead ECG, as measured during screening.
6. History of alcohol abuse at any time in life or history of other substance abuse within the past year, according to PI's assessment.
7. Significant hearing or visual impairment that may affect the patient's ability to complete the test procedures.
8. Concurrent major psychiatric condition (eg, major depressive disorder, schizophrenia, or bipolar disorder) as confirmed by the PI. Patients with additional diagnosis of autism spectrum disorder or anxiety disorder will be allowed.
9. Subject has active diseases that would interfere with participation, such as acquired immunodeficiency disorder, hepatitis C, hepatitis B, or tuberculosis.
10. Subject is planning to commence psychotherapy or CBT within 4 weeks prior to screening.
11. Patient is an immediate family member of anyone employed by the sponsor, PI, or study staff.
12. Patient has weight < 25 kg or a BMI greater than the 97th percentile for his age according to the Centers for Disease Control and Prevention (refer to Appendix 1). To participate in the Part 1 cohort receiving 50 mg dose, patient must weigh ≥ 75 lbs (34 kg).
13. Patient has participated in another clinical trial within the 30 days before screening.

    -

Ages: 9 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 163 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
NIH Toolbox Cognitive Battery cognition crystallized composite score | 13 Weeks
  The change from baseline to Week 13 in the NIH Toolbox Cognitive Battery cognition crystallized composite score (NIH-TCB CCC), which is calculated from the Picture Vocabulary and Oral Reading domains.

SECONDARY OUTCOMES:
NRS patient-specific behaviors within the domains of Daily Function, Language, and Academic Skills. | 13 Weeks
  Change from baseline to Week 13 in Numerical rating scale (NRS) scores based on patient-specific behaviors within the domains of Daily Function, Language, and Academic Skills.
CaGI-I for the general domains of Daily Function, Language, and Academic Skills. | 13 Weeks
  Change from baseline to Week 13 Caregiver Global Impression of Improvement (CaGI-I) for the general domains of Daily Function, Language, and Academic Skills.
Investigator rated (CGI-I) for the general domains of Daily Function, Language, and Academic Skills | 13 Weeks
  Change from baseline to Week 13 Clinical Global Impression Improvement - Investigator rated (CGI-I) for the general domains of Daily Function, Language, and Academic Skills
NRS scores based on patient-specific behaviors within the domain of Emotions/Behaviors | 13 Weeks
  Change from baseline to Week 13 NRS scores based on patient-specific behaviors within the domain of Emotions/Behaviors
CaGI-I for the general domain of Emotions/Behaviors | 13 Weeks
  Change from baseline to Week 13 CaGI-I for the general domain of Emotions/Behaviors
The NIH-TCB domains of Picture Vocabulary, Oral Reading Recognition, and Pattern Comparison Processing Speed | 13 Weeks
  Change from baseline to Week 13 the NIH-TCB domains of Picture Vocabulary, Oral Reading Recognition, and Pattern Comparison Processing Speed
Vineland-3 Adaptive Behavior Scale (Vineland-3) | 13 Weeks
  Change from baseline to Week 13 Vineland-3 Adaptive Behavior Scale (Vineland-3)
Verbal Knowledge test from the Stanford Binet (ed 5) (SB-5) IQ assessment | 13 Weeks
  Change from baseline Verbal Knowledge test from the Stanford Binet (ed 5) (SB-5) IQ assessment

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Amnova Clinical Research, Irvine, California
  - Thompson Autism & Neurodevelopment Center - CHOC, Orange, California
  - UC Davis, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - U Mass, Worcester, Massachusetts
  - Icahn School of Medicine at Mount Sinai Hospital, New York, New York
  - Cincinatti Children's Hospital Medical Center, Cincinnati, Ohio
  - Suburban Research Associates, Media, Pennsylvania
  - Clinic for Special Children, Strasburg, Pennsylvania
  - Greenwood Genetic Center, Greenville, South Carolina
  - University of Utah and Primary Childrens Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No